CLINICAL TRIAL: NCT04397575
Title: Cohorte Non Interventionnelle Ambispective Nationale Multicentrique de Patients Suivis Pour Cancer et infectés Par le SARS-CoV-2
Brief Title: The GCO-002 CACOVID-19 Cohort: a French Nationwide Multicenter Study of COVID-19 Infected Cancer Patients
Acronym: CACOVID-19
Status: Completed | Type: Observational
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other); GORTEC (Other); Intergroupe Francophone de Cancerologie Thoracique (Other); Association de Neuro-Oncologues d'Expression Francaise (Other)
Responsible Party: Sponsor
Other Study IDs: GCO002 CACOVID-19
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cancer; COVID; Solid Tumor; Social Inequality; French National Cohort; Chemotherapy; Immunotherapy; Surgery; Radiotherapy
Keywords: cancer; COVID; solid tumor; social inequality; french national cohort; chemotherapy; Immunotherapy; surgery; radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since December 2019, China and then the rest of the world have been affected by the rapid development of a new coronavirus, SARS-CoV-2 (severe acute respiratory syndrome corona virus 2). The disease caused by this coronavirus (COVID-19), which is transmitted by air via droplets, is potentially responsible for a severe respiratory syndrome but also for a multivisceral deficiency that can lead to death.

Cancer patients are generally more susceptible to infections than people without cancer due to immunosuppression caused by their tumor disease and/or conventional anti-cancer treatments used such as cytotoxic chemotherapy, several targeted therapies, radiotherapy or recent surgery. These patients may therefore be at particular risk for COVID-19.

This is suggested by the very first analysis on the subject, which reports data from the Chinese prospective database of 2007 patients with proven COVID-19 infection in 575 hospitals in 31 Chinese provinces. The authors of this publication conclude with 3 measures to be proposed to patients undergoing cancer follow-up: 1/ consider postponing adjuvant chemotherapy or surgery in the case of localized and stable cancer, 2/ reinforce protective measures for these patients, and 3/ monitor very closely and treat these patients more intensively when they have a COVID-19.

However, the increased risk of SARS-CoV-2 infection and severe forms of COVID-19 in cancer patients suggested by this first study remains to be demonstrated given its limitations, already highlighted by other authors. Indeed, the number of patients is small and the population of cancer patients is very heterogeneous, with in particular 12 patients out of 16 who had recovered from initial cancer treatments (therefore without immunosuppression), half of whom had a disease course of more than 4 years.

Nevertheless, a second Chinese study has just recently been published, reporting COVID-19 data among 1524 cancer patients admitted between December 30, 2019 and February 17, 2020 in the Department of Radiotherapy and Medical Oncology of the University Hospital of Wuhan, the source city of the COVID-19 epidemic. Although the rate of CoV-2 SARS infection was lower than that reported in the first study, it was still 0.79% (n=12), which is much higher than the rate of COVID-19 diagnosed in Wuhan City during the same period (0.37%, 41 152/11 081 000). Again, lung cancer was the main tumour location observed in 7 patients (58%), of which 5 (42%) were undergoing chemotherapy +/- immunotherapy. Three deaths (25%) were reported. Patients over 60 years of age with lung cancer had a higher incidence of COVID-19 (4.3% vs. 1.8%). Thus, it appears that the risk of COVID-19 is actually increased in cancer patients, although again, less than half of the patients with lung cancer had a higher incidence of COVID-19.

Moreover, two more recent studies performed in patients treated in Hubei Province of China and in New-York city found that patients with cancer had significantly increased risk of death compared to non-cancer COVID-19 patients, especially patients with metastatic cancer and those who had recent surgery.

Therefore, many questions remain to date on the level of risk and the severity of COVID-19 in patients with active cancer, in particular those under anti-cancer treatment and in patients recently operated for localized cancer.

DETAILED DESCRIPTION:
Since December 2019, China and then the rest of the world have been affected by the rapid development of a new coronavirus, SARS-CoV-2 (severe acute respiratory syndrome corona virus 2). The disease caused by this coronavirus (COVID-19), which is transmitted by air via droplets, is potentially responsible for a severe respiratory syndrome but also for a multivisceral deficiency that can lead to death.

In less than 3 months, the COVID-19 epidemic has already affected more than 440,000 persons and has been responsible for more than 20,000 deaths worldwide.

Cancer patients are generally more susceptible to infections than people without cancer due to immunosuppression caused by their tumor disease and/or conventional anti-cancer treatments used such as cytotoxic chemotherapy, several targeted therapies, radiotherapy or recent surgery. These patients may therefore be at particular risk for COVID-19.

This is suggested by the very first analysis on the subject, which reports data from the Chinese prospective database of 2007 patients with proven COVID-19 infection in 575 hospitals in 31 Chinese provinces. After exclusion of 417 cases without sufficient available clinical data, 1590 cases of patients infected with COVID-19 were analysed, of which 18 (1%) had a personal history of cancer. This prevalence was higher than that of COVID-19 in the general Chinese population since the beginning of the epidemic (0.29%). Lung cancer (n=5, 28%) and colorectal cancer (n=5, 28%) were the 2 most common cancers. Four (25%) of the 16 patients for whom treatment was known had received chemotherapy or had surgery in the month prior to COVID-19 infection, while the majority (n=12, 75%) were patients in remission or cured of their cancer after primary surgery. Compared to patients without cancer, patients with cancer were older (63 years vs. 48 years) and had a more frequent history of smoking (22% vs. 7%). Most importantly, patients with cancer had more severe forms of COVID-19 than patients without cancer (7/18 or 39% vs. 124/1572 or 8%, p=0.0003). Patients who had chemotherapy or surgery in the month preceding the diagnosis of COVID-19 had a significantly increased risk of the severe form (3/4 or 75% vs. 6/14 or 43%), which was confirmed in multivariate analysis after adjustment on other risk factors such as age, smoking and other comorbidities, with a relative risk of 5.34 (95% CI: 1.80-16.18;p=0.0026). Finally, patients with cancer deteriorated more rapidly than patients without cancer (13 days vs. 43 days, p<0.0001). The authors of this publication conclude with 3 measures to be proposed to patients undergoing cancer follow-up: 1/ consider postponing adjuvant chemotherapy or surgery in the case of localized and stable cancer, 2/ reinforce protective measures for these patients, and 3/ monitor very closely and treat these patients more intensively when they have a COVID-19.

However, the increased risk of SARS-CoV-2 infection and severe forms of COVID-19 in cancer patients suggested by this first study remains to be demonstrated given its limitations, already highlighted by other authors. Indeed, the number of patients is small and the population of cancer patients is very heterogeneous, with in particular 12 patients out of 16 who had recovered from initial cancer treatments (therefore without immunosuppression), half of whom had a disease course of more than 4 years.

Nevertheless, a second Chinese study has just recently been published, reporting COVID-19 data among 1524 cancer patients admitted between December 30, 2019 and February 17, 2020 in the Department of Radiotherapy and Medical Oncology of the University Hospital of Wuhan, the source city of the COVID-19 epidemic. Although the rate of CoV-2 SARS infection was lower than that reported in the first study, it was still 0.79% (n=12), which is much higher than the rate of COVID-19 diagnosed in Wuhan City during the same period (0.37%, 41 152/11 081 000). Again, lung cancer was the main tumor location observed in 7 patients (58%), of which 5 (42%) were undergoing chemotherapy +/- immunotherapy. Three deaths (25%) were reported. Patients over 60 years of age with lung cancer had a higher incidence of COVID-19 (4.3% vs. 1.8%). Thus, it appears that the risk of COVID-19 is actually increased in cancer patients, although again, less than half of the patients with lung cancer had a higher incidence of COVID-19.

Moreover, two more recent studies performed in patients treated in Hubei Province of China and in New-York city found that patients with cancer had significantly increased risk of death compared to non-cancer COVID-19 patients, especially patients with metastatic cancer and those who had recent surgery.

Therefore, many questions remain to date on the level of risk and the severity of COVID-19 in patients with active cancer, in particular those under anti-cancer treatment and in patients recently operated for localized cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient undergoing treatment or under surveillance or recently diagnosed and who has not yet started treatment for cancer at one of the following locations : digestive (esophagus, stomach, colorectal, small intestine, pancreas, biliary tract, Vater's ampulla, liver, GIST, neuroendocrine tumour, anal canal, primary peritoneum, appendix), thoracic (non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), mesothelioma), head and neck (oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, salivary glands, sinus), gynecological (breast, ovary, cervix, endometrium, vulva), central nervous system, dermatological, urological (prostate, kidney, bladder and upper urinary tract, external genitals)
* Patient with PCR and/or serology and/or CT-scan confirmed SARS-COV-2 infection or with suggestive COVID-19 syndrome (fever, fatigue, body aches, headache, cough, dyspnea, sudden onset of anosmia or ageusia in the absence of rhinitis or nasal obstruction) without biological or CT-scan confirmation during the period of March 1, 2020 to September 30, 2020.
* Inpatient or outpatient
* Patient informed of the research and, by way of derogation, patient treated in an emergency situation

Exclusion Criteria:

* Patients whose cancer in the cohort was treated curatively more than 5 years ago, with no evidence of recurrence at the time of the SARS-COV-2 infection.
* Patient expressing opposition to participating in the cohort
* Patient subject to a protective measure (patient under guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing treatment or under surveillance or recently diagnosed and who has not yet started treatment for cancer at one of the following locations : digestive (esophagus, stomach, colorectal, small intestine, pancreas, biliary tract, Vater's ampulla, liver, GIST, neuroendocrine tumour, anal canal, primary peritoneum, appendix), thoracic (non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), mesothelioma), head and neck (oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, salivary glands, sinus), gynecological (breast, ovary, cervix, endometrium, vulva), central nervous system, dermatological, urological (prostate, kidney, bladder and upper urinary tract, external genitals)
Sampling Method: Non-Probability Sample
Enrollment: 1523 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of cases of SARS-COV-2 infection and mortality rate directly related to the infection in patients being followed for digestive, thoracic, head and neck, gynecologic, cerebral, urologic or cutaneous cancer | 3 months
  Describe the number of cases of SARS-COV-2 infection, including those with severe form, and the mortality rate directly related to the infection in patients being followed for any of the following cancers: digestive, thoracic, head and neck, gynecologic, cerebral, urologic, or cutaneous

SECONDARY OUTCOMES:
Number of cases of SARS-COV-2 infection | 3 months
  Describe the number of cases of SARS-COV-2 infection according to:
  * Tumor location
  * metastatic or localized status
  * status treated or under surveillance
  * the type of cancer treatment n the 3 months prior to the occurrence of COVID-19 or more
Percentage of severe and fatal forms.of cases of SARS-COV-2 infection | 3 months
  Describe the percentage of severe and fatal forms respectively according to :
  * Tumor location
  * metastatic or localized status
  * status treated or under surveillance
  * type of cancer treatment received in the 3 months prior to the occurrence of COVID-19 or more
Social characteristics of individuals on treatment | 3 months
  Social characteristics of individuals (dwelling place with a INSE code, ) impact on the treatment management of cancer. Information of dwelling place (INSE code), socio-professional leve (INSEE classification) will be collected
Link between socio-territorial determinants and the characteristics/severity of SARS-COV-2 infection. | 3 months
  Analyze the link between socio-territorial determinants and the characteristics/severity of SARS-COV-2 infection, as well as the impact of the infection on cancer management.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile GIRAULT, Study Director — Federation Francophone de Cancerologie Digestive
Locations (148):
- France (148):
  - Ch D'Abbeville, Abbeville
  - CHU - Hôpital Sud, Amiens
  - CHU - Hôtel Dieu, Angers
  - Hôpital Privé, Antony
  - CH Victor Dupouy, Argenteuil
  - CH - Metz Thionville Mercy, Ars-Laquenexy
  - Hôpital Général d'Auch, Auch
  - Ch-Ght Unyon Auxerre, Auxerre
  - CH - Henri Duffaut, Avignon
  - PRIVE - Sainte Catherine, Avignon
  - CH, Bayeux
  - CH - Côte Basque, Bayonne
  - CH, Beauvais
  - CHU - Jean Minjoz, Besançon
  - PRIVE - Franche Comté, Besançon
  - PRIVE - Centre Pierre Curie, Beuvry
  - CH - Germon et Gauthier - Service de Gastroentérologie, Béthune
  - CH, Béziers
  - CH, Blois
  - PRIVE - Tivoli, Bordeaux
  - CHU - Ambroise Paré, Boulogne
  - CH - Duchenne, Boulogne-sur-Mer
  - CH - Fleyriat, Bourg-en-Bresse
  - CHU - Morvan, Brest
  - CHU - Pierre Wertheimer, Bron
  - CHU - Côte de Nacre, Caen
  - PRIVE - François Baclesse, Caen
  - CH, Calais
  - PRIVE - Infirmerie protestante, Caluire-et-Cuire
  - CH, Cannes
  - PRIVE - Médipole de Savoie, Challes-les-Eaux
  - PRIVE - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - CH, Charleville-Mézières
  - CH, Chauny
  - CH, Châlons-en-Champagne
  - CHP du Cotentin, Cherbourg
  - CH, Cholet
  - CH - HIA Percy, Clamart
  - CHU - Estaing, Clermont-Ferrand
  - PRIVE - CAC Jean PERRIN, Clermont-Ferrand
  - CHU - Beaujon, Clichy
  - CH - Hôpitaux civils de Colmar, Colmar
  - CHU - Louis MOURIER, Colombes
  - CH - Compiegne, Compiègne
  - PRIVE - Saint Côme, Compiègne
  - CH - Sud Francilien, Corbeil-Essonnes
  - PRIVE - Cédres, Cornebarrieu
  - PRIVE - Clinique de Flandre, Coudekerque-Branche
  - CH - GHPSO Site de Creil, Creil
  - Ch - C.H.I.C., Créteil
  - CHU - Henri Mondor, Créteil
  - PRIVE - Centre Léonard de Vinci, Dechy
  - CHU - Hôpital François Mitterand, Dijon
  - PRIVE - CAC GF Leclerc, Dijon
  - PRIVE - Institut de Cancérologie de Bourgogne GRReCC, Dijon
  - CH - Louis Pasteur, Dole
  - CH, Douai
  - CH - Victor Jousselin, Dreux
  - PRIVE - Clinique Claude Bernard, Ermont
  - PRIVE - Forcilles, Férolles-Attilly
  - CH - Frejus Saint Raphael, Fréjus
  - CH, Grasse
  - CHU - Grenoble Alpes, Grenoble
  - PRIVE - GHM Daniel Hollard, Grenoble
  - CH - Marne La Vallée/Jossigny, Jossigny
  - CH - CHD Vendée, La Roche-sur-Yon
  - CH - Louis Pasteur, Le Coudray
  - PRIVE - L'Estuaire, Le Havre
  - PRIVE - Centre Jean Bernard, Le Mans
  - CH - Docteur Schaffner, Lens
  - PRIVE - Teissier, Liévin
  - CH - Saint Vincent, Lille
  - CHU - Claude Huriez, Lille
  - PRIVE - CAC Oscar Lambret, Lille
  - PRIVE - La Louvière Institut de Cancérologie Lille Métropole, Lille
  - CH - Robert Bisson, Lisieux
  - CH - GH Nord Essone, Longjumeau
  - CH - CHBS Hôpital du Scrorff, Lorient
  - CHU - Edouard Herriot, Lyon
  - CHU - La Croix Rousse, Lyon
  - PRIVE - La Sauvegarde Lyon, Lyon
  - CH - La Conception, Marseille
  - CH - Saint Joseph, Marseille
  - CHU - La Timone, Marseille
  - CH - Les Chanaux, Mâcon
  - CH - GHI de l'Est Francilien Site de Meaux, Meaux
  - CH - Layné, Mont-de-Marsan
  - CH - Site du Mittan, Montbéliard
  - CH, Montélimar
  - CH - Emile Muller, Mulhouse
  - PRIVE - Oncologie Gentilly, Nancy
  - PRIVE - Confluent SAS, Nantes
  - PRIVE - Hartmann, Neuilly-sur-Seine
  - CH - Pierre Beregovoy, Nevers
  - CH, Niort
  - CHU - Caremeau, Nîmes
  - CHR - Centre Hospitalier Régional La Source, Orléans
  - AP - HP - Pitié Salpêtrière, Paris
  - Bichat, Paris
  - CHU - Cochin, Paris
  - CHU - Lariboisière, Paris
  - CHU - Saint Antoine, Paris
  - CHU - Saint Louis, Paris
  - CHU - Tenon, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - PRIVE - Saint Joseph, Paris
  - Privé - Montsouris, Paris
  - PRIVE - Centre Oncologie Catalan, Perpignan
  - CHU - Haut Lévêque, Pessac
  - CH, Périgueux
  - CHU - Lyon Sud, Pierre-Bénite
  - PRIVE - Centre Cario HPCA, Plérin
  - CHU - La Miletrie, Poitiers
  - CH - René Dubos, Pontoise
  - PRIVE - Clinique La Croix du Sud, Quint-Fonsegrives
  - CHU - Robert Debré, Reims
  - PRIVE - Polyclinique Courlancy, Reims
  - PRIVEE - Jean Godinot, Reims
  - PRIVEE - Polyclinique Courlancy, Reims
  - CHU - Charles Nicolle, Rouen
  - CAC - Institut Curie R. Huguenin, Saint-Cloud
  - PRIVE - Ramsay Sainte Loire, Saint-Etienne
  - PRIVE - Saint Grégoire, Saint-Grégoire
  - CH - Begin, Saint-Mandé
  - PRIVE - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU - Hôpital Nord CHU Saint Etienne, Saint-Priest-en-Jarez
  - PRIVE - Trenel, Sainte-Colombe
  - CH - Centre Hospitalier de Saint Malo, St-Malo
  - CHU - Hautepierre, Strasbourg
  - ICAN - Institut de Cancérologie de Strasbourg Europe, Strasbourg
  - PRIVE - Strasbourg Oncologie Libérale, Strasbourg
  - CH - Foch, Suresnes
  - CH - Maison Santé Protestante, Talence
  - CH - Birgorre, Tarbes
  - CH - Leman, Thonon-les-Bains
  - CH - Sainte Musse, Toulon
  - CAC - Oncopole, Toulouse
  - CHU - Rangueil, Toulouse
  - CH - Gustave Dron, Tourcoing
  - CHU - Bretonneau, Tours
  - CH, Valence
  - CH, Valenciennes
  - PRIVE - Dentellières, Valenciennes
  - CHU - Brabois, Vandœuvre-lès-Nancy
  - PRIVE - Robert Schuman, Vantoux
  - CH - Paul Morel, Vesoul
  - CAC - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study results — https://doi.org/10.1016/j.ejca.2020.09.035